CLINICAL TRIAL: NCT02247154
Title: A Study of the Safety and Efficacy of an Intravenous Immunoglobulin (Vigam® Liquid) in Patients With Primary or Secondary Antibody Deficiency.
Brief Title: A Study of the Safety and Efficacy of Vigam® Liquid in Patients With Primary or Secondary Antibody Deficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: VIGPSAD
Record Dates: First submitted 2014-09-02; First posted 2014-09-23 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Primary or Secondary Antibody Deficiency
MeSH Terms: interventions — gamma-Globulins

ARMS (1):
- Vigam® Liquid (Experimental)
  Interventions: Biological: Vigam® (Human Normal Immunoglobulin)

INTERVENTIONS:
Biological: Vigam® (Human Normal Immunoglobulin)

SUMMARY:
To determine:

1. The safety of Vigam® Liquid in patients with primary or secondary antibody deficiency (PAD or SAD).
2. The efficacy of Vigam® Liquid in patients with primary or secondary antibody deficiency.
3. The half-life of Vigam® Liquid after 4 months of treatment.
4. The subclass and total gammaglobulin concentrations after each infusion of Vigam® Liquid.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-80 years) with PAD or SAD
* With a low serum IgG (<6 g/l) and a history of recurrent infections
* Requiring and eligible for polyvalent intravenous immunoglobulin (IVIG) replacement therapy
* Non-reactive for HBsAg and with an alanine aminotransferase (ALT) level less than twice upper limit of normal prior to entry into the trial

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Primary Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
IgG half-life | Pre-dose, 5 min, 1, 2, 4, 7, 10, 14, 21 days post-dose

CONTACTS AND LOCATIONS:
Locations (8):
- United Kingdom (8):
  - Papworth Hospital, Papworth Everard, Cambridgeshire
  - Cardiff Royal Infirmary, Cardiff
  - Leicester Royal Infirmary, Leicester
  - Royal Brompton Hospital, London
  - Royal Free Hospital, London
  - Royal Victoria Infirmary, Newcastle
  - Hospital of St Cross, Rugby
  - Taunton & Somerset Hospital, Somerset

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk